CLINICAL TRIAL: NCT04982744
Title: Registry of Li Fraumeni and Li Fraumeni Like Syndromes That Collects Clinical, Functional, Genetic, Genealogical, Imaging, Surgical, Treatment, Quality of Life Data. Data is Linked to Patients' Biological Samples, When Available
Brief Title: Registry of Li Fraumeni and Li Fraumeni Like Syndromes
Acronym: ReLF
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Luca Sangiorgi, Head of Department of Rare Skeletal Disorders, Istituto Ortopedico Rizzoli
Other Study IDs: 579/2020/Oss/IOR
Record Dates: First submitted 2021-06-30; First posted 2021-07-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Li-Fraumeni Syndrome; Li-Fraumeni-Like Syndrome
Keywords: Disease Registry; Natural History Study; Genotype-Phenotype Correlation; Disease Evolution
MeSH Terms: conditions — Li-Fraumeni Syndrome; Li-Fraumeni-Like Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected by Li Fraumeni and Li Fraumeni Like syndromes: The group comprises all patients affected by Li Fraumeni and Li Fraumeni Like syndromes

SUMMARY:
ReLF is a retrospective and prospective registry, finalized for care and research purposes. It is articulated in main sections - strongly related and mutually dependent on each other - corresponding to different data domains: personal information, clinical data, genetic data, genealogical data, surgeries, etc. This approach has been developed to corroborate and integrate data from different resources and aspects of the diseases and to correlate genetic background and phenotypic outcomes, in order to better investigate diseases pathophysiology. Due to legal requirements, institutional directives and organizational issues, we are unable to include individuals residing outside Italy in the registry at this time. We are currently engaged in the preparation of a recruitment process for individuals residing outside Italy.

DETAILED DESCRIPTION:
The traditional method of collecting patient information is often chaotic, inconvenient, and sometimes even unsafe, particularly when dealing with rare diseases. In 2020, the need to simplify the diagnostic process and to overcome the difficulties of data storage and analysis, led to the suggestion of implementing the Registry of Li Fraumeni and Li Fraumeni Like syndromes (ReLF).

The ReLF relies on an IT Platform named GeDI (Genotype-phenotype Data Integration platform). This solution, realized by a collaboration among Department of Rare Skeletal Disorders and a local software-house (Dilaxia Spa), is a GDPR-compliant, multi-client, web-accessible system and it has been designed according to current medical informatics standards (Orphacode, ICD-10, Human Genome Variants Society, Findability Accessibility Interoperability Reusability -FAIR- Principles). GeDI is continuously implemented to improve management of persons with Li Fraumeni and Li Fraumeni Like Syndromes and to help researchers in analyzing collected information. ReLF is articulated in main sections:

* Personal data: it comprises general information, birth details and residence data;
* Patient data: including the patients internal code, the hospital code and other patient details;
* Diagnostic Process: the diagnosis, the status (affected, suspected, etc.), age at diagnosis, comorbidities, allergies, etc.;
* Genogram: a tool for designing the family transmission of the disease, alongside information on the disease status of all relatives included;
* Clinical events: it records a long list of signs and symptoms as well as several additional items to describe the disease
* Genetic Analysis and Alteration: including analytical technique, sample information, analysis duration, etc. This section also comprises detailed information on any detected pathological variants (e.g. gene, international reference, DNA change, protein change, genomic position, etc.);
* Visits: this section includes visit type (genetic, orthopedic, rehabilitation, pediatric, etc.), the date of the visit, prescriptions, imaging, etc.;
* Treatments: this section comprises information of a wide range of treatments including pharmacological, devices, supplements, and other treatments such as psychological, nutritional, etc.;
* Surgeries: this section contains information on the type of surgeries, the age of the patients, the site/localization of the procedures, etc.
* Documents: this repository allow us to store all types of documents (radiological reports, imaging, consents, clinical reports, etc.);
* Consents: this section provides a comprehensive overview of all consents collected, including the collection date;
* Samples: this section includes information on the samples, like the type, date of collection, etc.
* PROs: this section collects information on patients reported outcomes such as the quality of life or ABC scale.

ELIGIBILITY:
Inclusion Criteria:

* All patients affected by Li Fraumeni or Li Fraumeni Like syndromes

Exclusion Criteria:

* Any condition unrelated to Li Fraumeni or Li Fraumeni Like syndromes

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by Li Fraumeni or Li Fraumeni Like syndromes
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2045-07 (Estimated)

PRIMARY OUTCOMES:
Natural History and Epidemiology | Since the disease is rare, the timeframe is strictly related to patients enrolment and consequently to amount of collected data. Considering the low prevalence of this disease, the time frame is up to 10 years.
  Assessment of epidemiological information. Anthropometric data: weight in kg, height in cm. In addition, weight and height will be combined to report BMI as kg/m^2 Clinical details of the tumor: site of the lesion, number of recurrence(s), presence/absence of metastasis, size of lesion in cm^3 Additional clinical data: type of surgery, age at surgery in years are updated at each follow up and retrospectively (when possible).
  Clinical reports, medical charts and imaging are the primary source of data.

SECONDARY OUTCOMES:
Genotype-Phenotype Correlation | The timeframe is strictly related to patients enrolment and consequently to amount of collected data. Considering the low prevalence of this disease, the time frame is up to 10 years.
  The secondary outcome comprises the correlation between genotype and phenotype. This includes, but is not limited to, clinical features and genetic background. This will be pursued using the information collected during visits and follow-ups and the genetic information resulting from molecular investigations.
  Collection of genetics background (target gene, type of mutation, clinical significance are reported following HGVS nomenclature) and family history (in terms of inheritance by maternal or paternal line).
  Anthropometric data (weight in kg, height in cm. In addition, weight and height will be combined to report BMI in kg/m^2), clinical details (site of the lesion, recurrence, metastasis), orthopedic and functional features are updated at each follow up.

OTHER OUTCOMES:
Inter- and intra-familial oncological characterization | The timeframe is strictly related to patients enrolment and consequently to amount of collected data. Considering the low prevalence of this disease, the time frame is up to 10 years.
  This outcome aims to investigate similarities and difference of tumoral manifestation (site of the tumor, type of tumor, age at onset, grade of lesion) in patients affected by Li Fraumeni or Li Fraumeni Like syndromes within the families and among the families.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Sangiorgi, MSc, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (2):
- Italy (2):
  - Irccs Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna
  - IRCCS Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna